CLINICAL TRIAL: NCT05858515
Title: REVERSE-Long COVID: A Multicenter Randomized, Placebo-Controlled Clinical Trial of Immunomodulation (With Baricitinib) for Long COVID Related Cognitive Impairment and ADRD (Alzheimer's Disease and Related Dementias)
Brief Title: REVERSE-Long COVID-19 With Baricitinib Study
Acronym: REVERSE-LC
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This submission for the pilot study has been withdrawn as the full trial opened under a different NCT number before participants enrolled in the pilot.
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Emory University (Other); University of California, San Francisco (Other); University of Minnesota (Other); Vanderbilt University (Other); Yale University (Other)
Responsible Party: Principal Investigator, Wes Ely, Co-Director, Critical Illness, Brain Dysfunction, and Survivorship Center, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: U13800
Record Dates: First submitted 2023-03-28; First posted 2023-05-15 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Post-Acute COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — baricitinib

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blind, parallel-design superiority design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The block size and treatment allocation will only be known to the biostatistician creating the randomization list and will not be shared with trial investigators or any other study personnel. This list will be directly uploaded into REDCap's randomization module. This maintains the concealment of future allocations and has been used successfully for several of our large RCTs. The details of the randomization procedure including details regarding stratification and block sizes will fully be reported in the trial publication to enable readers to assess the risk of bias. Randomization assignments will be accessible 24 hours a day, 7 days a week to the study coordinators and staff
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): These participants will receive placebo for 24 weeks (6 mo)
  Interventions: Drug: Placebo
- Intervention #1 (Experimental): These participants will receive baricitinib 4 mg daily for 24 weeks
  Interventions: Drug: Baricitinib 4 MG

INTERVENTIONS:
Drug: Baricitinib 4 MG — Nonproprietary name: Baricitinib
  Other Names: Olumiant
  Arms: Intervention #1
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
REVERSE-LC is a phase 3 trial of baricitinib versus placebo in adults with neurocognitive impairment (a form of Alzheimer's Disease and Related Dementias or ADRD) or cardiopulmonary symptoms due to Long COVID.

DETAILED DESCRIPTION:
This is a multi-site randomized, placebo-controlled, double-blind, parallel-design REVERSE-LC phase 3 study. Individuals meeting inclusion criteria will be randomized to one of two arms: the intervention arm of baricitinib 4 mg daily for 24 weeks (dose adjusted to 2 mg or 1 mg for baseline renal dysfunction) versus the placebo arm for 24 weeks. In addition to safety, a variety of clinical and biological outcome measures will be assessed.

ELIGIBILITY:
In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Obtain a signed and dated informed consent form from participant
2. State their willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged ≥18 years old
4. Meet the following criteria for "Post-COVID Condition" or Long COVID:

   1. 6-months prior, documented SARS-CoV-2 infection
   2. Cognitive impairment as defined by having at least 20% positive (worse or much worse) items on the ECOG assessment
   3. Neurocognitive symptoms must have been present for at least 60 days prior to screening. Symptoms that wax and wane must have been initially present at least 60 days prior to screening.
5. Ability to take oral medication and be willing to adhere to the baricitinib regimen
6. Females of childbearing potential must agree to either abstinence or use at least one acceptable method of contraception from the time of screening though at least 28 days after the end of the study intervention period. Note: Acceptable methods include barrier contraceptives (condoms or diaphragm) with spermicide, intrauterine devices (IUDs), hormonal contraceptives, oral contraceptive pills, and surgical sterilization.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pre-existing cognitive impairment not exacerbated by acute COVID as determined by study physicians after thorough review of participant's history and medical records
2. Current use of baricitinib or other disease-modifying antirheumatic drug (DMARDs)
3. Known allergic reactions to components of the baricitinib
4. Have ever been randomized in this study or any other study investigating baricitinib
5. Positive SARS-CoV-2 PCR or rapid Antigen test in the past 14 days
6. Pregnancy or breastfeeding
7. Any history of venous thromboembolism ever
8. History of malignancy or lymphoproliferative disorder
9. Renal dysfunction with estimated glomerular filtration rate of < 30 mL/min/1.73m2
10. Absolute Neutrophil Count (ANC) <1200 cells/mm3
11. History or evidence of severe or end-stage liver disease (e.g. bilirubin ≥1.5x or AST/ALT >2x normal).
12. Positive Hepatitis B surface antibody, antigen or core antibody, or Positive Hepatitis C RNR or antigen
13. Positive HIV 4th generation (antibody/antigen) ELISA test
14. Have had symptomatic herpes zoster infection within 3 months prior to study entry or have a history of disseminated/complicated herpes zoster or herpes simplex infection
15. History of latent (diagnosed with Quantiferon testing) or active tuberculosis
16. History of a current or recent (< 30 days from screening) clinically significant viral, bacterial, fungal, or parasitic infection
17. History of chronic alcohol abuse, Intravenous (IV) drug abuse, or other illicit drug abuse within the 2 years prior to study entry
18. Are immunocompromised and, in the opinion of the investigator, are at an unacceptable risk for participating in the study
19. Treatment with another investigational drug or other intervention < 30 days of study enrollment
20. Are unable or unwilling to make themselves available for the duration of the study and/or are unwilling to follow study restrictions/procedures
21. Severe cognitive, physical, or psychological disability that would prevent participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Enrollment | 6 months
  2 participants per month, on average, are randomized
Diversity in enrollment | 6 months
  40% of participants will be from individuals disproportionally affected by COVID (Black, Hispanic, Asian, American Indian)
Study drug prescribed | 9 months
  80% of participants received every prescribed dose of the study drug
Study withdrawals | 18 months
  Less than 20% participants will be deemed lost to follow up
Adverse event reporting | 18 months
  100% of Serious Adverse Events reported to Data Safety Monitoring Board within 24 hours of study team awareness
Study dosing | 9 months
  100% adherence to study drug dose adjustments guidelines
Study completion | 18 months
  80% of participants adhere to all study procedures and requirements

SECONDARY OUTCOMES:
Severe and Serious Adverse Events | 9 months
  Compare the percentage of severe and serious adverse events between study arms from baseline to week 12.
Premature study discontinuation | 9 months
  Compare the rate of study drug/placebo premature discontinuation by study arm (tolerability)
Global Neuropsychological Function | 9 months
  Assess percentage changes of global neuropsychological function as measured using the CNS Vital Signs Neurocognition Index cognitive battery between baricitinib and placebo study arm from baseline to week 12.
Cardiopulmonary testing | 9 months
  Assess percentage changes of exercise capacity (peak VO2) using cardiopulmonary exercise testing (CPET) in the baricitinib arm compared to the placebo arm from baseline to week 12
Everyday Cognition | 9 months
  Assess percentage changes of cognitive impairment using Everyday Cognition (ECog) scale in the baricitinib arm compared to the placebo arm from baseline to week 12
Functional Status | 9 months
  Assess percentage changes of functional status measures in the baricitinib arm compared to the placebo arm from baseline to week 12
Quality of Life Measures | 9 months
  Assess percentage changes of quality of life measures in the baricitinib arm compared to the placebo arm from baseline to week 12
Post-Exertional Malaise | 9 months
  Assess percentage changes of post-exertional malaise using De Paul Symptom Questionnaire - Post-Exertional Malaise (DSQ-PEM) in the baricitinib arm compared to the placebo arm from baseline to week 12
Shortness of Breath | 9 months
  Assess percentage changes of the effect of breathlessness on daily activities using the Modified Medical Research Council Dyspnea Scale (mMRC) in the baricitinib arm compared to the placebo arm from baseline to week 12
Symptom Burden | 9 months
  Assess percentage changes of post COVID-19 symptom burden using the Symptom Burden Questionnaire for Long COVID (SBQ-LC) Circulation Subscale in the baricitinib arm compared to the placebo arm from baseline to week 12
Inflammation biomarkers | 9 months
  Decreases in plasma biomarkers of inflammation in the baricitinib arm compared to placebo arm from baseline to week 12
Viral Reservoirs | 9 months
  Decreases in viral reservoirs for the baricitinib arm compared to placebo arm from baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: E. Wesley Ely, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (6):
- United States (6):
  - University of California San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Emory University, Atlanta, Georgia
  - University of Minnesota, Minneapolis, Minnesota
  - Vanderbilt University, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee